CLINICAL TRIAL: NCT05258903
Title: Ulnar Artery Versus Radial Artery Cannulation in Paediatric Patients: a Prospective Randomized Non-inferiority Study
Brief Title: Ulnar Artery Versus Radial Artery Cannulation in Paediatric Patients
Acronym: ULNART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KDAR FN Brno Artery
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arterial Catheterization
Keywords: pediatric anesthesia; pediatric patient; Arterial catheterization; arterial catheter; ultrasound-guided cannulation; Arterial cannulation

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: randomization after general anesthesia induction, or deep sedation in PICU
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulnar artery (Experimental): Ulnar artery cannulation under USG-guidance
  Interventions: Procedure: Ulnar artery cannulation
- Radial artery (Active Comparator): Radial artery cannulation under USG-guidance
  Interventions: Procedure: Radial artery cannulation

INTERVENTIONS:
Procedure: Ulnar artery cannulation — Ulnar artery will be cannulated under USG guidance
  Other Names: Ulnar artery catheterization
  Arms: Ulnar artery
Procedure: Radial artery cannulation — Radial artery will be cannulated under USG guidance
  Other Names: Radial artery catheterization
  Arms: Radial artery

SUMMARY:
Arterial cannulation is indicated in several clinical settings: high-risk surgery, respiratory failure, circulatory failure. The possible anatomical sites of cannulation are: a.radialis, a.brachialis, a. femoralis. However, the most reported complications in preschool-aged children are associated with femoral and brachial arteries. Therefore, alternative cannulation sites are being searched as ulnar artery, tibial posterior artery.

DETAILED DESCRIPTION:
In pediatric patients, artery cannulation may be associated with a higher risk of complications. The preferred puncture site is the radial artery or the femoral artery. However, puncture of the femoral artery in comparison with the radial artery is based on observational data as a significant risk side of post-puncture complications. The radial artery is the dominant artery of the hand, and the collateral supply (via the ulnar artery) is often unable to provide adequate peripheral perfusion. Therefore, other potential sites suitable for artery cannulation in paediatric patients are currently being investigated with the primary goal of increasing safety and reducing the risk of post-puncture complications. According to published studies, the potential alternatives are: posterior tibial artery and ulnar artery. Both arteries have comparable dimensions with radial artery and can be used for USG-guided cannulation. In this prospective randomized trial, patients with clinical indication for arterial cannulation (high-risk surgery, respiratory failure, circulatory failure) undergoing surgery under general anesthesia and pediatric patients admitted into the pediatric intensive care unit (PICU) will be randomized in form of sealed envelopes into a.radialis and a.ulnaris group as the initial site of arterial catheterization. Ultrasound (USG) measurement of both arteries will be performed before the cannulation. The catheterization success rate (number of percutaneous punctures) and overall success rate will be evaluated. The artery will be cannulated under USG control, initially in in-plane view, only in case of insufficient image, or after 2 unsuccessful attempts, the out-of-plane approach could be used. The maximum 5 percutaneous attempts and 10 minutes could be used for the initial (randomized) site of cannulation). In case of cannulation failure, the other artery could be used for cannulation. The rate of complications in 24 hours after cannulation will be evaluated. The arterial catheter will stay in place until the clinical indication remained.

.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients (1 - 6 years)
* high risk surgery (significant blood loss or hemodynamic instability)
* critically ill patients at PICU (respiratory failure, circulatory failure)
* informed consent

Exclusion Criteria:

* refused to participate
* arterial catheterization not clinically relevant

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
overall puncture success in different arterial sites | intraoperatively
  defined by number of required percutaneous punctures and overall site success rate

SECONDARY OUTCOMES:
Arteries anatomical description | intraoperatively
  Defined by USG measurement of depth of the artery - (distance from the skin to the upper wall of the artery), cross-sectional area, diameter of the artery.
Technique of the ultrasound-guided cannulation (in-plane/out-of-plane) | intraoperatively
  The USG guidance approach will be evaluated
Incidence of complications | 24 hours postoperatively
  Blood supply disorder, trophic changes, hematoma, arterial wall injury (aneurysm etc.), thrombosis.
Duration of catheterization | Intraoperatively
  Time needed for successful catheterization
Interval between catheterization and catheter removal | 24 hours postoperatively
  Interval between catheterization and catheter removal will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided